CLINICAL TRIAL: NCT04889651
Title: A Randomized, Open Label, Single Dose, Full Replicated Crossover Study to Compare the Pharmacokinetics and Safety Between BR9004 and BR9004-1 in Healthy Male Volunteers
Brief Title: A Study to Compare the Pharmacokinetics and Safety Between BR9004 and BR9004-1 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-ABT-CT-101
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(TRTR) (Experimental): The selected subjects are randomized into two sequence group(Sequence A (TRTR) & Sequence B (RTRT)).
  * Sequence A: T-R-T-R
  * T: BR9004, oral single-dose administration, 1 tablet per day
  * R: BR9004-1, oral single-dose administration, 1 tablet per day
  * Washout interval between periods: 7 days
  Interventions: Drug: BR9004; Drug: BR9004-1
- B(RTRT) (Experimental): The selected subjects are randomized into two sequence group(Sequence A (TRTR) & Sequence B (RTRT)).
  * Sequence B: R-T-R-T
  * T: BR9004, oral single-dose administration, 1 tablet per day
  * R: BR9004-1, oral single-dose administration, 1 tablet per day
  * Washout interval between periods: 7 days
  Interventions: Drug: BR9004; Drug: BR9004-1

INTERVENTIONS:
Drug: BR9004 — BR9004: Abiraterone acetate 200mg, Boryung Pharmaceutical Co., Ltd.
  Other Names: Abiraterone acetate 200mg
Drug: BR9004-1 — BR9004-1: Zytiga Tab. 500mg (Abiraterone acetate 500mg), Janssen Korea
  Other Names: Zytiga Tab

SUMMARY:
To compare the pharmacokinetics and safety between BR9004 and BR9004-1 in healthy male subjects after a single-dose administration while fasting.

DETAILED DESCRIPTION:
This is a randomized, open label, single dose, full replicated crossover study to compare the pharmacokinetics and safety between BR9004 and BR9004-1 in healthy male subjects under fasting conditions. To this end, subjects were divided into two sequence groups [Sequence A (TRTR) & Sequence B (RTRT), T: BR9004, single oral administration, R: BR9004-1, single oral administration].

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily signed the Institutional Review Board(IRB)-approved informed consent to participate in this study after being given an sufficient explanation about the study objectives, details, and characteristics of the investigational product
2. Healthy males aged between 19 and 55 at the time of the screening test
3. Those who weigh over 50 kg with BMI of 18.0 to 30.0 BMI (kg/m2) = Weight(kg) / [Height(m)]2

Exclusion Criteria:

1. Those who had a clinically significant medical history such as hypersensitivity reaction, intolerance, and anaphylaxis against Abiraterone which is the main ingredient of the investigational products.
2. Those who had clinically significant diseases in the liver, kidneys, digestive, respiratory, musculoskeletal, endocrine, neuropsychiatric, hematologic, oncologic, and cardiovascular disorders (including orthostatic hypotension), etc.
3. Those who had gastrointestinal disorders (e.g., Crohn's disease, ulcerative colitis, etc.) that may affect the absorption of the investigational products or underwent surgeries (excluding appendectomy, hernia surgery, endoscopic removal of polys, and surgeries for piles, anal fissure, anal fistula)
4. Those who were judged to have clinically significant abnormal results in the interview, vital signs, ECG, physical examinations, blood & urine test, etc. during the screening test
5. Those who showed positive results in HBsAg, hepatitis C virus(HCV) Ab, HIV Ab, and rapid plasma reagin(RPR) test during the screening test
6. Those who showed one of the following results during the screening test:

   * Aspartate aminotransferase(AST) or Alanine aminotransferase(ALT) higher than 2 times the upper limit of normal range
   * T. bilirubin higher than 2 times than the upper limit of normal range
   * Estimated Glomerular Filtration Rate(e-GFR) lower than 60 mL/min/1.73m2 (using the Chronic Kidney Disease Epidemiology Collaboration(CKD-EPI))
7. Those who showed > 150 mmHg or < 90 mmHg of systolic blood pressure or > 95 mmHg or < 60 mmHg of diastolic blood pressure during the screening test
8. Those who did not agree to stop taking prohibited drugs (prescription drugs, over-the-counter drugs, herbal medicines or nutritional supplements, e.g., vitamins) within 2 weeks after the administration of investigational products (accepted if the investigator judges that the drug may not affect the safety of the subject and study results)
9. Those who had drug abuse (especially drugs that affect the central nervous system such as sleeping pills, analgesics that work on the central nervous system(CNS), narcotic drugs, or psychoactive drugs) or have a history of drug abuse
10. Those who had a continuous intake of alcohol that exceeds 21 units/week (1 unit=10g=12.5mL) within 6 months of the screening

    ☞ Amount of alcohol(g) = Amount of intake (ml) x Alcohol degree (%) x 0.8* (*10g=12.5mL)
11. Those who smoked over 10 cigarettes a day within 6 months of the screening
12. Those administered with the investigational products by participating in other clinical studies within 180 days before the first administration of the investigational products (however, the day after the last administration date is considered Day 1 after the previous study participation ends)
13. Those who donated whole blood within 8 weeks and plasma or platelet within 4 weeks before the first administration of the investigational products or who did not agree to stop donating blood donation for 30 days from the date when the investigational products are administered
14. Those who did not agree to stop having foods diets (especially those containing grape fruit-containing foods) that may affect the absorption, distribution, metabolism, and excretion of the investigational products from 3 days before the first administration until the last visit
15. Those who did not agree to use clinically accepted contraceptive methods (e.g., contraceptive pills, intrauterine devices, sterilization procedures(vasectomy, and tubal ligation) or barrier methods (combined use of spermicide and condom, contraceptive diaphragm, vaginal sponge or cervical cap)) for at least 3 weeks after the last administration from the first administration of investigational products.
16. Those who have genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption, etc.
17. Those undergoing combined therapy with radium-223 chloride
18. Those whom the investigator judges unsuitable for participation in this study for other reasons

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables-Cmax | 1~22 days after medication
  Maximum observed plasma concentration(Cmax) of BR9004 and BR9004-1
Pharmacokinetic variables-AUClast | 1~22 days after medication
  Area under the plasma drug concentration-time curve over the time interval from 0 to the last quantifiable plasma concentration(AUClast) of BR9004 and BR9004-1

SECONDARY OUTCOMES:
Pharmacokinetic variables-t1/2β | 1~22 days after medication
  Terminal half-life(t1/2β) of BR9004 and BR9004-1
Pharmacokinetic variables-Tmax | 1~22 days after medication
  Time of maximum concentration(Tmax) of BR9004 and BR9004-1
Pharmacokinetic variables-AUCinf | 1~22 days after medication
  Area under the plasma drug concentration-time curve over the time interval from 0 to extrapolated to infinity(AUCinf) of BR9004 and BR9004-1

CONTACTS AND LOCATIONS:
Overall Officials: An-Hye Kim, Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Gyeonggi-do, Seongnam-si, South Korea